CLINICAL TRIAL: NCT07205159
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Safety and Efficacy of FB102 in Patients With Severe to Very Severe Alopecia Areata.
Brief Title: A Study to Evaluate the Safety and Efficacy of FB102 in Patients With Severe to Very Severe Alopecia Areata.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Forte Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FB102-701
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB102 (Active Comparator): Participants will receive FB102.
  Interventions: Drug: FB102
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB102 — Route of administration- Intravenous (IV)
  Arms: FB102
Drug: Placebo — Route of administration- Intravenous (IV)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of FB102 in patients with severe to very severe alopecia areata (AA).

DETAILED DESCRIPTION:
Up to approximately 32 participants who meet all the Screening eligibility criteria will be randomized in a 3:1 ratio to receive FB102, or placebo dosing to match.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-60 years and females aged 18-75 years at Screening.
* Clinical diagnosis of severe to very severe AA with ≥50% scalp hair loss (including AT or AU) confirmed by SALT score and central photo review; no other cause of hair loss.

  * AT = complete scalp hair loss; AU = complete scalp, facial, and body hair loss. Note: There are additional inclusion criteria. The study center will determine if participant meets all of the criteria

Exclusion Criteria:

* Other types of alopecia (e.g., diffuse AA, traction, scarring alopecia, telogen effluvium, trichotillomania, chemotherapy-induced hair loss, androgenetic alopecia).
* Other scalp diseases impacting AA assessment (e.g., psoriasis, dermatitis, tinea capitis).
* Active systemic diseases causing hair loss (e.g., lupus, thyroiditis, systemic sclerosis, lichen planus, syphilis).

Note: There are additional exclusion criteria. The study center will determine if participant meets all of the criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Upto 36 Weeks post first dose administration
Change from Baseline of Severity of Alopecia Tool (SALT) score at Week 16. | From Screening through Week 16.
  The Severity of Alopecia Tool (SALT) score ranges from 0 (no scalp hair loss) to 100 (complete scalp hair loss), with higher scores indicating greater severity. Change from baseline in SALT score at Week 16 will assess treatment effect. The AA-IGA categorizes SALT scores as follows: 0 = None (0%), 1 = Limited (1-20%), 2 = Moderate (21-49%), 3 = Severe (50-94%), 4 = Very Severe (95-100%).

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - St Leonards, Saint Leonards, New South Wales (nsw)
  - Coorparoo, Coorparoo, Queensland
  - South Yarra, South Yarra, Victoria
- New Zealand (3):
  - Auckland, Auckland, Auckland
  - Christchurch, Christchurch, Canterbury
  - Palmerston North, Palmerston North, Palmerston North Central